CLINICAL TRIAL: NCT05824273
Title: Leveraging Social Media to Increase Lung Cancer Screening Awareness, Knowledge and Uptake in High-Risk Populations
Brief Title: The INSPIRE-Lung Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pro2022-0860; 7R01CA263662-02 (NIH)
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
Keywords: Lung cancer screening; Social media; Tailored interventions
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored health communication intervention (LungTalk) (Experimental): Participants will receive the tailored health intervention "LungTalk". LungTalk is a 10-15 minute long computer-tailored health communication and decision-making tool that is theoretically grounded in the Conceptual Model on Lung Cancer Screening Participation.
  Interventions: Behavioral: LungTalk
- Non-tailored Intervention (Active Comparator): Participants will receive non-tailored American Cancer Society (ACS) Lung Screening Informational Video as per standard of care. ACS Lung Screening Informational Video (ACS LSIV) is a non-tailored 5-minute video from the American Cancer Society about lung cancer screening designed for the lay individual.
  Interventions: Behavioral: Non-tailored intervention - Standard of practice

INTERVENTIONS:
Behavioral: LungTalk — LungTalk is a 10-15 minute long computer-tailored health communication and decision-making tool.
  Arms: Tailored health communication intervention (LungTalk)
Behavioral: Non-tailored intervention - Standard of practice — ACS Lung Screening Informational Video
  Arms: Non-tailored Intervention

SUMMARY:
LungTalk and leveraging Facebook-targeted Advertisement (FBTA) addresses the call to develop and test multi-level, cancer communication interventions using innovative methods and designs. The study's long term goal is to increase lung cancer screening uptake among appropriate, high-risk individuals nationwide.

ELIGIBILITY:
Inclusion Criteria:

* ≥20-pack-year smoking history;
* Individuals who currently smoke or quit smoking within the past 15 years

Exclusion Criteria:

* Previously undergone LDCT for early detection of lung cancer, have a lung nodule or nodules that are currently being followed
* Has ever been diagnosed with lung cancer
* Individuals with impaired decision-making (because our primary outcome is decision-making, we will not include individuals with impaired decision-making)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carter-Bawa, PhD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Meridian Health - Center for Discovery and Innovation, Nutley, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Final recommendation statement: Lung cancer screening. U. S. Preventive Services Task Force. Updated March 9, 2021. Accessed May 26, 2021, 2021. https://www.uspreventiveservicestaskforce.org/uspstf/document/RecommendationStatementFinal/lung-cancer-screening
- [Background] United States Preventive Services Task Force. Final recommendation statement: Lung cancer screening. Updated Updated December 2016. Accessed May 21, 2020. http://www.uspreventiveservicestaskforce.org/Page/Document/RecommendationStatementFinal/lung-cancer-screening
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] De Koning H. ES 02.01 The Dutch-Belgian Lung Cancer Screening Trial (NELSON). Journal of Thoracic Oncology. 2017;12(11):S1611. doi:10.1016/j.jtho.2017.09.108
- [Background] Centers for Medicare & Medicaid Services. Decision memo for screening for lung cancer with low-dose computed tomography (LDCT) (CAG-00439N). Accessed May 21, 2020. https://www.cms.gov/medicare-coverage-database/details/nca-decision-memo.aspx?NCAId=274
- [Background] Okereke IC, Nishi S, Zhou J, Goodwin JS. Trends in lung cancer screening in the United States, 2016-2017. J Thorac Dis. 2019 Mar;11(3):873-881. doi: 10.21037/jtd.2019.01.105. PMID 31019776
- [Background] Carter-Harris L, Ceppa DP, Hanna N, Rawl SM. Lung cancer screening: what do long-term smokers know and believe? Health Expect. 2017 Feb;20(1):59-68. doi: 10.1111/hex.12433. Epub 2015 Dec 23. PMID 26701339
- [Background] Carter-Harris L, Brandzel S, Wernli KJ, Roth JA, Buist DSM. A qualitative study exploring why individuals opt out of lung cancer screening. Fam Pract. 2017 Apr 1;34(2):239-244. doi: 10.1093/fampra/cmw146. PMID 28122849
- [Background] Carter-Harris L, Slaven JE Jr, Monahan PO, Shedd-Steele R, Hanna N, Rawl SM. Understanding lung cancer screening behavior: Racial, gender, and geographic differences among Indiana long-term smokers. Prev Med Rep. 2018 Feb 3;10:49-54. doi: 10.1016/j.pmedr.2018.01.018. eCollection 2018 Jun. PMID 29552458
- [Background] Carter-Harris L, Comer RS, Goyal A, Vode EC, Hanna N, Ceppa D, Rawl SM. Development and Usability Testing of a Computer-Tailored Decision Support Tool for Lung Cancer Screening: Study Protocol. JMIR Res Protoc. 2017 Nov 16;6(11):e225. doi: 10.2196/resprot.8694. PMID 29146565
- [Background] Chambers DA, Glasgow RE, Stange KC. The dynamic sustainability framework: addressing the paradox of sustainment amid ongoing change. Implement Sci. 2013 Oct 2;8:117. doi: 10.1186/1748-5908-8-117. PMID 24088228
- [Background] United States Preventive Services Task Force. Final recommendation statement: Lung cancer screening. Accessed October 10. http://www.uspreventiveservicestaskforce.org/Page/Document/RecommendationStatementFinal/lung-cancer-screening
- [Background] United States Preventive Services Task Force. Draft recommendation statement: lung cancer: Screening July 7, 2020. Accessed October 10. https://uspreventiveservicestaskforce.org/uspstf/draft-recommendation/lung-cancer-screening-2020
- [Background] Carter-Harris L, Comer RS, Slaven Ii JE, Monahan PO, Vode E, Hanna NH, Ceppa DP, Rawl SM. Computer-Tailored Decision Support Tool for Lung Cancer Screening: Community-Based Pilot Randomized Controlled Trial. J Med Internet Res. 2020 Nov 3;22(11):e17050. doi: 10.2196/17050. PMID 33141096
- [Background] Carter-Harris L, Tan AS, Salloum RG, Young-Wolff KC. Patient-provider discussions about lung cancer screening pre- and post-guidelines: Health Information National Trends Survey (HINTS). Patient Educ Couns. 2016 Nov;99(11):1772-1777. doi: 10.1016/j.pec.2016.05.014. Epub 2016 May 17. PMID 27241830
- [Background] Carter-Harris L, Slaven JE 2nd, Monohan P, Rawl SM. Development and Psychometric Evaluation of the Lung Cancer Screening Health Belief Scales. Cancer Nurs. 2017 May/Jun;40(3):237-244. doi: 10.1097/NCC.0000000000000386. PMID 27244666
- [Background] Carter-Harris L, Slaven JE 2nd, Monahan PO, Draucker CB, Vode E, Rawl SM. Understanding lung cancer screening behaviour using path analysis. J Med Screen. 2020 Jun;27(2):105-112. doi: 10.1177/0969141319876961. Epub 2019 Sep 24. PMID 31550991
- [Background] Carter-Harris L, Bartlett Ellis R, Warrick A, Rawl S. Beyond Traditional Newspaper Advertisement: Leveraging Facebook-Targeted Advertisement to Recruit Long-Term Smokers for Research. J Med Internet Res. 2016 Jun 15;18(6):e117. doi: 10.2196/jmir.5502. PMID 27306780
- [Background] Facebook Distribution of Users by Age Group in the U.S. Facebook. Accessed May 26, 2021, 2021. https://www.statista.com/statistics/187549/facebook-distribution-of-users-age-group-usa/
- [Background] Frandsen M, Walters J, Ferguson SG. Exploring the viability of using online social media advertising as a recruitment method for smoking cessation clinical trials. Nicotine Tob Res. 2014 Feb;16(2):247-51. doi: 10.1093/ntr/ntt157. Epub 2013 Oct 14. PMID 24127266
- [Background] Ramo DE, Prochaska JJ. Broad reach and targeted recruitment using Facebook for an online survey of young adult substance use. J Med Internet Res. 2012 Feb 23;14(1):e28. doi: 10.2196/jmir.1878. PMID 22360969
- [Background] Ramo DE, Hall SM, Prochaska JJ. Reaching young adult smokers through the internet: comparison of three recruitment mechanisms. Nicotine Tob Res. 2010 Jul;12(7):768-75. doi: 10.1093/ntr/ntq086. Epub 2010 Jun 7. PMID 20530194
- [Background] Ramo DE, Delucchi KL, Liu H, Hall SM, Prochaska JJ. Young adults who smoke cigarettes and marijuana: analysis of thoughts and behaviors. Addict Behav. 2014 Jan;39(1):77-84. doi: 10.1016/j.addbeh.2013.08.035. Epub 2013 Sep 7. PMID 24090626
- [Background] Smith A, Anderson M. Social media use in 2018. Pew Internet.org. Updated October 9. https://www.pewinternet.org/2018/03/01/social-media-use-in-2018/
- [Background] United States Adults Social Platform Use. Social networking platforms' demographics update 2019. Marketingcharts.com,. Accessed October 9, https://www.marketingcharts.com/charts/us-adults-social-platform-use-demographic-group-2019/attachment/pew-social-platform-use-by-demographic-apr2019
- [Background] Albada A, Ausems MG, Bensing JM, van Dulmen S. Tailored information about cancer risk and screening: a systematic review. Patient Educ Couns. 2009 Nov;77(2):155-71. doi: 10.1016/j.pec.2009.03.005. Epub 2009 Apr 18. PMID 19376676
- [Background] Krebs P, Prochaska JO, Rossi JS. A meta-analysis of computer-tailored interventions for health behavior change. Prev Med. 2010 Sep-Oct;51(3-4):214-21. doi: 10.1016/j.ypmed.2010.06.004. Epub 2010 Jun 15. PMID 20558196
- [Background] Noar SM, Benac CN, Harris MS. Does tailoring matter? Meta-analytic review of tailored print health behavior change interventions. Psychol Bull. 2007 Jul;133(4):673-93. doi: 10.1037/0033-2909.133.4.673. PMID 17592961
- [Background] Kreuter M, Farrell D, Olevitch L, Brennan L. Tailoring health messages: Customizing communication with computer technology. Tailoring health messages: Customizing communication with computer technology. Lawrence Erlbaum Associates Publishers; 2000:xiii, 270-xiii, 270.
- [Background] Rawl SM, Skinner CS, Perkins SM, Springston J, Wang HL, Russell KM, Tong Y, Gebregziabher N, Krier C, Smith-Howell E, Brady-Watts T, Myers LJ, Ballard D, Rhyant B, Willis DR, Imperiale TF, Champion VL. Computer-delivered tailored intervention improves colon cancer screening knowledge and health beliefs of African-Americans. Health Educ Res. 2012 Oct;27(5):868-85. doi: 10.1093/her/cys094. Epub 2012 Aug 27. PMID 22926008
- [Background] Ruffin MT 4th, Fetters MD, Jimbo M. Preference-based electronic decision aid to promote colorectal cancer screening: results of a randomized controlled trial. Prev Med. 2007 Oct;45(4):267-73. doi: 10.1016/j.ypmed.2007.07.003. Epub 2007 Jul 14. PMID 17689600
- [Background] Wu TY, Lin C. Developing and evaluating an individually tailored intervention to increase mammography adherence among Chinese American women. Cancer Nurs. 2015 Jan-Feb;38(1):40-9. doi: 10.1097/NCC.0000000000000126. PMID 24621965
- [Background] Ahmad F, Cameron JI, Stewart DE. A tailored intervention to promote breast cancer screening among South Asian immigrant women. Soc Sci Med. 2005 Feb;60(3):575-86. doi: 10.1016/j.socscimed.2004.05.018. PMID 15550305
- [Background] Champion V, Foster JL, Menon U. Tailoring interventions for health behavior change in breast cancer screening. Cancer Pract. 1997 Sep-Oct;5(5):283-8. PMID 9341350
- [Background] Lau YK, Caverly TJ, Cherng ST, Cao P, West M, Arenberg D, Meza R. Development and validation of a personalized, web-based decision aid for lung cancer screening using mixed methods: a study protocol. JMIR Res Protoc. 2014 Dec 19;3(4):e78. doi: 10.2196/resprot.4039. PMID 25532218
- [Background] Memorial Sloan Kettering Cancer Center. Memorial Sloan Kettering Cancer Center, Lung cancer screening decision tool. Accessibility verified February 12, 2016. Accessed October 7, 2020. http://nomograms.mskcc.org/Lung/Screening.aspx
- [Background] Chen Y, Marcus MW, Niaz A, Duffy SW, Field JK. My Lung Risk: a user-friendly, web-based calculator for risk assessment of lung cancer based on the validated Liverpool Lung Project risk prediction model. International Journal of Health Promotion and Education. 2014/05/04 2014;52(3):144-152. doi:10.1080/14635240.2014.888814
- [Background] Volk RJ, Linder SK, Leal VB, Rabius V, Cinciripini PM, Kamath GR, Munden RF, Bevers TB. Feasibility of a patient decision aid about lung cancer screening with low-dose computed tomography. Prev Med. 2014 May;62:60-3. doi: 10.1016/j.ypmed.2014.02.006. Epub 2014 Feb 8. PMID 24518006
- [Background] Veterans Health Administration. Veterans Health Administration, Screening for lung cancer pamphlet. Accessibility verified February 12, 2016. Accessed September 29,. http://www.prevention.va.gov/docs/LungCancerScreeningHandout.pdf.
- [Background] Dharod A, Bellinger C, Foley K, Case LD, Miller D. The Reach and Feasibility of an Interactive Lung Cancer Screening Decision Aid Delivered by Patient Portal. Appl Clin Inform. 2019 Jan;10(1):19-27. doi: 10.1055/s-0038-1676807. Epub 2019 Jan 9. PMID 30625501
- [Background] Carter-Harris L, Davis LL, Rawl SM. Lung Cancer Screening Participation: Developing a Conceptual Model to Guide Research. Res Theory Nurs Pract. 2016 Nov 1;30(4):333-352. doi: 10.1891/1541-6577.30.4.333. PMID 28304262
- [Background] McDonnell KK, Strayer SM, Sercy E, Campbell C, Friedman DB, Cartmell KB, Eberth JM. Developing and testing a brief clinic-based lung cancer screening decision aid for primary care settings. Health Expect. 2018 Aug;21(4):796-804. doi: 10.1111/hex.12675. Epub 2018 Feb 23. PMID 29473696
- [Background] American Cancer Society. Cancer Screening Tests Videos. Accessed October 9. https://www.cancer.org/healthy/find-cancer-early/cancer-screening-tests-videos.html
- [Background] American Cancer Society. Lung Cancer Screening Guidelines. Accessed October 9. https://www.cancer.org/health-care-professionals/american-cancer-society-prevention-early-detection-guidelines/lung-cancer-screening-guidelines.html
- [Background] FACEBOOK for developers. Facebook Analytics Accessed October 9, 2020. https://developers.facebook.com/docs/analytics/
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Russomanno J, Patterson JG, Jabson Tree JM. Social Media Recruitment of Marginalized, Hard-to-Reach Populations: Development of Recruitment and Monitoring Guidelines. JMIR Public Health Surveill. 2019 Dec 2;5(4):e14886. doi: 10.2196/14886. PMID 31789598
- [Background] GO2 Foundation. Screening Centers of Excellence citation. Accessed October 9, 2020, (https://go2foundation.org/risk-early-detection/screening-centers/)
- [Background] Raudenbush Stephen W, Bryk Anthony S, eds. Hierarchical Linear Models: Applications and Data Analysis Methods. 2 ed. SAGE Publications, Inc.; 2002.
- [Background] Graham JW, Hofer SM, Donaldson SI, MacKinnon DP, Schafer JL. Analysis with missing data in prevention research. In: Bryant K, Windle M, West S, eds. The science of prevention: methodological advances from alcohol and substance abuse research. American Psychological Association; 1997:325-366.
- [Background] Schafer JL, Olsen MK. Multiple Imputation for Multivariate Missing-Data Problems: A Data Analyst's Perspective. Multivariate Behav Res. 1998 Oct 1;33(4):545-71. doi: 10.1207/s15327906mbr3304_5. PMID 26753828
- [Background] Hedeker D, Gibbons RD. Application of random-effects pattern-mixture models for missing data in longitudinal studies. Psychological Methods. 1997;2(1):64-78. doi:10.1037/1082-989X.2.1.64
- [Background] Benjamini Y, Hochberg Y. On the Adaptive Control of the False Discovery Rate in Multiple Testing With Independent Statistics. Journal of Educational and Behavioral Statistics. 2000;25(1):60-83. doi:10.3102/10769986025001060
- [Background] Arigo D, Pagoto S, Carter-Harris L, Lillie SE, Nebeker C. Using social media for health research: Methodological and ethical considerations for recruitment and intervention delivery. Digit Health. 2018 May 7;4:2055207618771757. doi: 10.1177/2055207618771757. eCollection 2018 Jan-Dec. PMID 29942634
- [Derived] Carter-Bawa L, Banerjee SC, Comer RS, Kale MS, King JC, Leopold KT, Monahan PO, Ostroff JS, Slaven JE Jr, Valenzona F, Wiener RS, Rawl SM. Leveraging social media to increase lung cancer screening awareness, knowledge and uptake among high-risk populations (The INSPIRE-Lung Study): study protocol of design and methods of a community-based randomized controlled trial. BMC Public Health. 2023 May 26;23(1):975. doi: 10.1186/s12889-023-15857-8. PMID 37237339
- [Derived] Lisa CB, Banerjee SC, Ostroff JS, Kale MS, King JC, Leopold KT, Monahan PO, Slaven JE Jr, Wiener RS, Valenzona F, Rawl SM, Comer RS. Leveraging social media to increase lung cancer screening awareness, knowledge and uptake among high-risk populations (The INSPIRE-Lung Study): Study protocol of design and methods of a community-based randomized controlled trial. Res Sq [Preprint]. 2023 May 4:rs.3.rs-2846041. doi: 10.21203/rs.3.rs-2846041/v1. PMID 37205569

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We initially had 512 participants enroll in the study. Still, only 483 were randomized to the study arms, as the remaining 29 participants were lost to follow-up after failing to complete the baseline survey upon enrollment.
Period: Overall Study
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Started | 256 | 256
Completed | 240 | 243
Not Completed | 16 | 13
Not completed — Lost to Follow-up | 16 | 13

BASELINE CHARACTERISTICS:
Population: Results are reported in aggregate because the baseline characteristics were collected prior to randomization, and there were no arm-specific differences at this stage.
Groups:
- Consented Patients to the Study: Results are reported in aggregate because the baseline characteristics were collected prior to randomization, and there were no arm-specific differences at this stage.
Arm/Group | Consented Patients to the Study
Number analyzed (Participants) | 483
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 269
  >=65 years | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (6.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 246
  Male | 236
  Non-binary | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 453
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 70
  White | 376
  More than one race | 7
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 483

OUTCOME MEASURES:

1. Primary Outcome: Reaching Screening Eligible Individuals Via Social Media - Reach
Description: Leveraging a well-established, social media-based platform (Facebook) to target screening-eligible individuals in the community. This will be measured by the total number of people who saw the FBTA at least once.
Time Frame: 11-month period ad remained active on Facebook
Population: Facebook-provided metrics were collected at the aggregate level (impressions, reach, engagements, and clicks). Because individual-level identifiers were not captured, it is not possible to report a precise 'number of people analyzed' from the platform; therefore, all Facebook-derived outcomes are reported as aggregate counts and rates. The total reach number on FB which is 3,109,482 is used instead.
Measure: Number; unit: participants
Groups:
- Unique Facebook Users Who Saw the Add: Number of unique Facebook users who saw the ad for the period of study recruitment.
Arm/Group | Unique Facebook Users Who Saw the Add
Number analyzed (Participants) | 3109482
participants | 1048191

2. Primary Outcome: Reaching Screening Eligible Individuals Via Social Media - Link Clicks
Description: Leveraging a well-established, social media-based platform (Facebook) to target screening-eligible individuals in the community. This will be measured by the total number of clicks on the link within the FBTA that led to the REDCap survey platform of the study.
Time Frame: 11-month period ad remained active on Facebook
Population: Overall Number of Participants Analyzed represents the number of participants screened for study interest prior to enrollment
Measure: Number; unit: unique clicks
Groups:
- Unique Facebook Users Who Clicked on the Link: Unique Facebook users who saw the ad and clicked on the link to be directed to the study-specific screening survey.
Arm/Group | Unique Facebook Users Who Clicked on the Link
Number analyzed (Participants) | 1048191
unique clicks | 24816

3. Primary Outcome: Reaching Screening Eligible Individuals Via Social Media - Impressions
Description: Leveraging a well-established, social media-based platform (Facebook) to target screening-eligible individuals in the community. This will be measured by the total number of times the FBTA was on screen (may include multiple views of the ad by the same person/people).
Time Frame: 11-month period ad remained active on Facebook
Population: as for outcome 1
Measure: Number; unit: number of times the add was viewed
Groups:
- Ad on Screen: Total number of times the ad was on Facebook screen during the study enrollment period.
Arm/Group | Ad on Screen
Number analyzed (Participants) | 3109482
number of times the add was viewed | 3109482

4. Primary Outcome: Effectiveness of LungTalk - Knowledge Assessment
Description: The assessment plan is intended to compare the effectiveness of a tailored (LungTalk) versus non-tailored health communication and decision support tool delivered online to improve total knowledge about lung screening. The total Knowledge of Lung Cancer Screening will be assessed with a 9-item multidimensional scale ranging from 0 to 9 with 0 being "No Knowledge" and 9 being "Complete knowledge".
Time Frame: At baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
score on a scale | 4 [0 to 9] | 4 [0 to 9]

5. Primary Outcome: Effectiveness of LungTalk - Knowledge Assessment
Description: as for outcome 4
Time Frame: At one week from baseline survey completion
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
score on a scale | 6 [1 to 9] | 6 [1 to 9]

6. Primary Outcome: Effectiveness of LungTalk - Perceived Risk
Description: The assessment plan is intended to compare the effectiveness of a tailored (LungTalk) versus non-tailored health communication and decision support tool delivered online to improve Perceived Risk. Perceived Risk of Lung Cancer is a 3-item scale with Likert-type responses. The range of scores is 3 to 12 (higher perceived risk of lung cancer).
Time Frame: At baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
score on a scale | 6 [3 to 12] | 6 [3 to 12]

7. Primary Outcome: Effectiveness of LungTalk - Perceived Risk
Description: as for outcome 6
Time Frame: At one week from baseline survey completion
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
score on a scale | 7 [3 to 12] | 7 [3 to 12]

8. Primary Outcome: Effectiveness of LungTalk - Perceived Benefits
Description: The assessment plan is intended to compare the effectiveness of a tailored (LungTalk) versus non-tailored health communication and decision support tool delivered online to improve Perceived Benefits. Perceived Benefits of Lung Cancer Screening is a 6-item scale with responses ranging from 1=strongly disagree to 4=strongly agree. The range of scores is 6 to 24 (higher perceived benefits).
Time Frame: At baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
score on a scale | 20 [6 to 24] | 19 [6 to 24]

9. Primary Outcome: Effectiveness of LungTalk - Perceived Benefits
Description: as for outcome 8
Time Frame: At one week from baseline survey completion
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
score on a scale | 20.5 [7 to 24] | 21 [6 to 24]

10. Primary Outcome: Effectiveness of LungTalk - Perceived Barriers
Description: The assessment plan is intended to compare the effectiveness of a tailored (LungTalk) versus non-tailored health communication and decision support tool delivered online to improve Perceived Barriers. Perceived Barriers to Lung Cancer Screening. This scale has 17 items with four-point Likert responses where 1=strongly disagree and 4=strongly agree. The range of scores is 17 to 68 (higher perceived barriers).
Time Frame: At baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
score on a scale | 33 [17 to 66] | 31 [17 to 68]

11. Primary Outcome: Effectiveness of LungTalk - Perceived Barriers
Description: as for outcome 10
Time Frame: At one week from baseline survey completion
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
score on a scale | 25 [17 to 58] | 25 [17 to 54]

12. Primary Outcome: Effectiveness of LungTalk - Self-Efficacy
Description: The assessment plan is intended to compare the effectiveness of a tailored (LungTalk) versus non-tailored health communication and decision support tool delivered online to improve Self-Efficacy. Self-Efficacy for Lung Cancer Screening will be assessed using a scale with nine items with a four-point Likert response option to assess individual beliefs about ability to arrange and complete a low-dose computed tomography (LDCT) to screen for lung cancer. The range of scores is 9 to 36 (higher levels of self-efficacy).
Time Frame: At baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
score on a scale | 31 [15 to 36] | 31 [15 to 36]

13. Primary Outcome: Effectiveness of LungTalk - Self-Efficacy
Description: as for outcome 12
Time Frame: At one week from baseline survey completion
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
score on a scale | 33 [14 to 36] | 33 [18 to 36]

14. Primary Outcome: Effectiveness of LungTalk - Occurrence of a Patient-Clinician Discussion
Description: The assessment plan is intended to compare the effectiveness of a tailored (LungTalk) versus non-tailored health communication and decision support tool delivered online to improve Occurrence of a Patient-Clinician Discussion. Occurrence of a Patient-Clinician Discussion about Lung Cancer Screening will be assessed with a single item requiring dichotomous (Y/N) response regarding a discussion with their healthcare provider.
Time Frame: At baseline
Population: The number of participants who reported having discussed with their health care provider regarding lung screening at any time prior to their enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
Participants | 91 | 92

15. Primary Outcome: Effectiveness of LungTalk - Occurrence of a Patient-Clinician Discussion
Description: as for outcome 14
Time Frame: At one week from baseline survey completion
Population: The number of participants who reported having discussed with their health care provider regarding lung screening since viewing the program.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
Participants | 113 | 115

16. Primary Outcome: Effectiveness of LungTalk - Occurrence of a Patient-Clinician Discussion
Description: as for outcome 14
Time Frame: At 6 months from baseline survey completion
Population: The number of participants who discussed with their health care provider about lung screening since viewing the program, captured at 6 months post survey completion.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 236 | 231
Participants | 193 | 161

17. Primary Outcome: Effectiveness of LungTalk - Screening Uptake
Description: The assessment plan is intended to compare the effectiveness of a tailored (LungTalk) versus non-tailored health communication and decision support tool delivered online to improve Screening Uptake, Lung Cancer Screening Uptake will be assessed via self-report via the stages of adoption algorithm for lung screening. There are seven stages (unaware, aware but unengaged, undecided, decided not to act, decided to act, action, and maintenance).
Time Frame: At baseline
Population: The number of participants who had a lung scan (low dose CAT scan) to screen for lung cancer prior to their enrolment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
Participants | 67 | 65

18. Primary Outcome: Effectiveness of LungTalk - Screening Uptake
Description: as for outcome 17
Time Frame: At one week from baseline survey completion
Population: The number of participants who had a lung scan (low dose CAT scan) to screen for lung cancer since joining this study (captured at 1 week post survey completion).
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 240 | 243
Participants | 48 | 45

19. Primary Outcome: Effectiveness of LungTalk - Screening Uptake
Description: as for outcome 17
Time Frame: At 6 months from baseline survey completion
Population: The number of participants who had a lung scan (low dose CAT scan) to screen for lung cancer since joining this study (captured at 6 months post baseline survey completion).
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
Number analyzed (Participants) | 236 | 231
Participants | 134 | 125

ADVERSE EVENTS:
Time Frame: 6 months post-enrolment for all participants who completed the baseline survey
Description: Any adverse events reported
Arm/Group | Tailored Health Communication Intervention (LungTalk) | Non-tailored Intervention
All-Cause Mortality (participants affected / at risk) | 0/240 | 0/243
Serious Adverse Events (participants affected / at risk) | 0/240 | 0/243
Other Adverse Events (participants affected / at risk) | 0/240 | 0/243

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT05824273/Prot_SAP_000.pdf